CLINICAL TRIAL: NCT02302781
Title: Why Subfertile Couples Drop Out (Drop Out Trial); a Prospective Survey in the Netherlands.
Brief Title: Why Subfertile Couples Drop Out
Acronym: DOT
Status: Completed | Type: Observational
Sponsor: Isala (Other)
Collaborators: Erasmus Medical Center (Other); Elisabeth-TweeSteden Ziekenhuis (Other); Reinier de Graaf Groep (Other); St. Antonius Hospital (Other); Maxima Medical Center (Other); Noordwest Ziekenhuisgroep (Other)
Responsible Party: Principal Investigator, B.J. Cohlen, Dr. B.J. Cohlen, Fertility Centre Isala, Isala
Other Study IDs: NL47393.075.14
Record Dates: First submitted 2014-11-25; First posted 2014-11-27 (Estimated); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Subfertility
Keywords: Reasons for Dropout; Subfertility; IVF; NON IVF
MeSH Terms: conditions — Infertility | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subfertile couples: Couples referred to one of the four participating hospitals with any type of subfertility for work up and/ or treatment will be screened for inclusion. Couples have not visited only other clinic yet.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Several validated questionnaires, depending on moment in fertility work up or treatment.

SUMMARY:
Dropout rates for fertility treatments are high. This study will examine the rate of patients that drop out during any type of subfertility work up or treatment. Furthermore, we will determine what reasons for discontinuation are and we will identify the demographic characteristics of the couples and the prognostic factors for drop out during assessment or treatment at a Fertility Centre in the Isala (Zwolle), Erasmus University Centre (Rotterdam), Elisabeth Twee Steden Hospital (Tilburg), Reinier de Graaf Group (Voorburg), St Antonius Hospital (Nieuwegein), Maxima Medical Centre (Veldhoven) and Noordwest Hospital Group (Den Helder/Alkmaar) in The Netherlands.

DETAILED DESCRIPTION:
Rationale Although fertility success rates are rising due to improved techniques and patients are usually highly motivated at their first visit of the clinic, dropout rates are high. Research has shown that fertility treatment is a cause for physical, psychological and economic burden.

Objective The aim of this study is to examine the rate of patient drop out during any type of subfertility work up or treatment. Furthermore, the investigators want to determine what the reasons for discontinuation are and to identify the demographic characteristics of these couples and the prognostic factors for drop out during assessment or treatment at a fertility clinic.

Study design Prospective cohort study at the fertility centres of Isala (Zwolle - The Netherlands), Erasmus University Centre (Rotterdam- The Netherlands), Elisabeth Twee Steden Hospital (Tilburg - The Netherlands), Reinier de Graaf Group (Voorburg - The Netherlands), St Antonius Hospital (Nieuwegein - The Netherlands), Maxima Medical Centre (Veldhoven - The Netherlands) and Noordwest Hospital Group (Den Helder/Alkmaar - The Netherlands).

Study population Every couple that undergoes any type of work up or treatment for subfertility problems and that has not visited any other clinic yet.

Methods Patient records of included couples will be studied and included patients will be asked to fill in a validated questionnaire after evaluations during work up or treatment. The data from both will be put in a database and analysed.

First visit (Q1) EPQ-RSS, SCREENIVF, MMQ, FertiQoL, demographic questions (128 items)

Evaluation (Q2) FertiQoL, HADS (48 items)

Evaluation (Q3) >4-6 cycles non-IVF (Q3) FertiQoL, HADS (48 items)

Evaluation (Q4) > 3 cycles IVF (Q4) FertiQoL, HADS (48 items)

Dropout (Q5) FertiQol, SCREENIVF, MMQ, PCQ-infertility, reasons for dropout (128 items)

Pregnancy (Q6) PCQ-infertility (53 items)

ELIGIBILITY:
Inclusion Criteria:

* Couples with any type of subfertility referred to one of the four participating centres
* Both partners are willing and able to separately fill out the questionnaires.

Exclusion Criteria:

* Unable to read or speak the Dutch language
* Medical contra-indication for pregnancy
* Previous OFO (initial infertility consultation), non IVF or IVF/ICSI cycles

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Couples referred to one of the four participating hospitals with any type of subfertility for work up and/ or treatment will be screened for inclusion. Couples have not visited any other clinic yet.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Dropout rates | 5 years
  To identify dropout rates at all stages of fertility care at the fertility centres of Isala (Zwolle), Erasmus MC (Rotterdam), IVF centre Voorburg (Voorburg), st Elisabeth (Tilburg).

SECONDARY OUTCOMES:
Reasons | 5 years
  Investigate the reasons for dropout, using the 'reason for dropout' questionnaire (made by the researchteam).
Patient satisfaction | 5 years
  Examine patient satisfaction with received fertility care, using the 'patient centredness questionnaire infertility' (PCQ-infertility).
Demographic characteristics | 5 years
  Identify demographic characteristics of dropout patients, using the 'demographic questions' (made by the researchteam).
Predictors | 5 years
  Identify predictors for discontinuation, using the 'Eysenck personality questionnaire' (short version or EPQ-RSS), the 'SCREENIVF' (including 'Hospital anxiety and depression scale' or HADS) questionnaire, the 'fertility quality of life questionnaire' (FertiQol) and the 'Maudsley Marital Questionnaire' (MMQ).

CONTACTS AND LOCATIONS:
Overall Officials: B.J. Cohlen, MD/PhD, Principal Investigator — Isala Zwolle
Locations (7):
- Netherlands (7):
  - Elisabeth Twee Stedeb Hospital, Tilburg, North Brabant
  - Maxima Medisch Centrum, Veldhoven, North Brabant
  - Noordwest Ziekenhuis Groep, Den Helder, North Holland
  - Isala, Zwolle, Overijssel
  - Erasmus Medical Centre, Rotterdam, South Holland
  - Reinier de Graaf Ziekenhuis Groep, Voorburg, South Holland
  - St Antonius Hospital, Nieuwegein, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aarts JW, van Empel IW, Boivin J, Nelen WL, Kremer JA, Verhaak CM. Relationship between quality of life and distress in infertility: a validation study of the Dutch FertiQoL. Hum Reprod. 2011 May;26(5):1112-8. doi: 10.1093/humrep/der051. Epub 2011 Mar 3. PMID 21372046
- [Background] Aarts JW, Huppelschoten AG, van Empel IW, Boivin J, Verhaak CM, Kremer JA, Nelen WL. How patient-centred care relates to patients' quality of life and distress: a study in 427 women experiencing infertility. Hum Reprod. 2012 Feb;27(2):488-95. doi: 10.1093/humrep/der386. Epub 2011 Nov 22. PMID 22108249
- [Background] Boivin J, Takefman J, Braverman A. The fertility quality of life (FertiQoL) tool: development and general psychometric properties. Hum Reprod. 2011 Aug;26(8):2084-91. doi: 10.1093/humrep/der171. Epub 2011 Jun 10. PMID 21665875
- [Background] Brandes M, van der Steen JO, Bokdam SB, Hamilton CJ, de Bruin JP, Nelen WL, Kremer JA. When and why do subfertile couples discontinue their fertility care? A longitudinal cohort study in a secondary care subfertility population. Hum Reprod. 2009 Dec;24(12):3127-35. doi: 10.1093/humrep/dep340. Epub 2009 Sep 26. PMID 19783833
- [Background] Dawson AA, Diedrich K, Felberbaum RE. Why do couples refuse or discontinue ART? Arch Gynecol Obstet. 2005 Nov;273(1):3-11. doi: 10.1007/s00404-005-0010-5. Epub 2005 Oct 28. PMID 16080011
- [Background] van Dongen AJ, Verhagen TE, Dumoulin JC, Land JA, Evers JL. Reasons for dropping out from a waiting list for in vitro fertilization. Fertil Steril. 2010 Oct;94(5):1713-6. doi: 10.1016/j.fertnstert.2009.08.066. Epub 2009 Nov 6. PMID 19896662
- [Background] van Empel IW, Aarts JW, Cohlen BJ, Huppelschoten DA, Laven JS, Nelen WL, Kremer JA. Measuring patient-centredness, the neglected outcome in fertility care: a random multicentre validation study. Hum Reprod. 2010 Oct;25(10):2516-26. doi: 10.1093/humrep/deq219. Epub 2010 Aug 18. PMID 20719811
- [Background] Gameiro S, Boivin J, Peronace L, Verhaak CM. Why do patients discontinue fertility treatment? A systematic review of reasons and predictors of discontinuation in fertility treatment. Hum Reprod Update. 2012 Nov-Dec;18(6):652-69. doi: 10.1093/humupd/dms031. Epub 2012 Aug 6. PMID 22869759
- [Background] Joseph O, Alfons V, Rob S. Further validation of the Maudsley Marital Questionnaire (MMQ). Psychol Health Med. 2007 May;12(3):346-52. doi: 10.1080/13548500600855481. PMID 17510905
- [Background] McDowell S, Murray A. Barriers to continuing in vitro fertilisation--why do patients exit fertility treatment? Aust N Z J Obstet Gynaecol. 2011 Feb;51(1):84-90. doi: 10.1111/j.1479-828X.2010.01236.x. Epub 2010 Oct 22. PMID 21299515
- [Background] Olivius C, Friden B, Borg G, Bergh C. Why do couples discontinue in vitro fertilization treatment? A cohort study. Fertil Steril. 2004 Feb;81(2):258-61. doi: 10.1016/j.fertnstert.2003.06.029. PMID 14967352
- [Background] Rajkhowa M, McConnell A, Thomas GE. Reasons for discontinuation of IVF treatment: a questionnaire study. Hum Reprod. 2006 Feb;21(2):358-63. doi: 10.1093/humrep/dei355. Epub 2005 Nov 3. PMID 16269448
- [Background] Smeenk JM, Verhaak CM, Stolwijk AM, Kremer JA, Braat DD. Reasons for dropout in an in vitro fertilization/intracytoplasmic sperm injection program. Fertil Steril. 2004 Feb;81(2):262-8. doi: 10.1016/j.fertnstert.2003.09.027. PMID 14967353
- [Background] Spinhoven P, Ormel J, Sloekers PP, Kempen GI, Speckens AE, Van Hemert AM. A validation study of the Hospital Anxiety and Depression Scale (HADS) in different groups of Dutch subjects. Psychol Med. 1997 Mar;27(2):363-70. doi: 10.1017/s0033291796004382. PMID 9089829
- [Background] Van den Broeck U, Holvoet L, Enzlin P, Bakelants E, Demyttenaere K, D'Hooghe T. Reasons for dropout in infertility treatment. Gynecol Obstet Invest. 2009;68(1):58-64. doi: 10.1159/000214839. Epub 2009 Apr 25. PMID 19401627
- [Background] Verberg MF, Eijkemans MJ, Heijnen EM, Broekmans FJ, de Klerk C, Fauser BC, Macklon NS. Why do couples drop-out from IVF treatment? A prospective cohort study. Hum Reprod. 2008 Sep;23(9):2050-5. doi: 10.1093/humrep/den219. Epub 2008 Jun 10. PMID 18544578
- [Background] Verhaak CM, Lintsen AM, Evers AW, Braat DD. Who is at risk of emotional problems and how do you know? Screening of women going for IVF treatment. Hum Reprod. 2010 May;25(5):1234-40. doi: 10.1093/humrep/deq054. Epub 2010 Mar 13. PMID 20228392
- [Background] Boivin J, Domar AD, Shapiro DB, Wischmann TH, Fauser BC, Verhaak C. Tackling burden in ART: an integrated approach for medical staff. Hum Reprod. 2012 Apr;27(4):941-50. doi: 10.1093/humrep/der467. Epub 2012 Jan 18. PMID 22258661
- [Background] Boivin J, Griffiths E, Venetis CA. Emotional distress in infertile women and failure of assisted reproductive technologies: meta-analysis of prospective psychosocial studies. BMJ. 2011 Feb 23;342:d223. doi: 10.1136/bmj.d223. PMID 21345903
- [Background] Boivin J, Lancastle D. Medical waiting periods: imminence, emotions and coping. Womens Health (Lond). 2010 Jan;6(1):59-69. doi: 10.2217/whe.09.79. PMID 20088730
- [Background] Sharma V, Allgar V, Rajkhowa M. Factors influencing the cumulative conception rate and discontinuation of in vitro fertilization treatment for infertility. Fertil Steril. 2002 Jul;78(1):40-6. doi: 10.1016/s0015-0282(02)03160-6. PMID 12095488
- [Background] Verhaak CM, Smeenk JM, Evers AW, Kremer JA, Kraaimaat FW, Braat DD. Women's emotional adjustment to IVF: a systematic review of 25 years of research. Hum Reprod Update. 2007 Jan-Feb;13(1):27-36. doi: 10.1093/humupd/dml040. Epub 2006 Aug 29. PMID 16940360